CLINICAL TRIAL: NCT06065865
Title: 'Effectively Intervening in Traumatized Parents and Children After Structural Domestic Violence: A Multiple Baseline Analysis'
Brief Title: 'Effectively Intervening in Traumatized Parents and Young Children After Structural Domestic Violence: A Multiple Baseline Analysis'
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Responsible Party: Principal Investigator, Lenneke Alink, Prof. dr., Universiteit Leiden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL84677.018.23
Record Dates: First submitted 2023-09-15; First posted 2023-10-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Domestic Violence; PTSD
Keywords: domestic violence; trauma; attachment; individualized treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The current study has a single case experimental design (SCED), more specifically, a non-concurrent multiple baseline design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guidance document (Experimental): The intervention that is investigated in this study is a guidance document, which is used to individualize the treatment trajectory for the parent-child dyad. This guidance document includes different factors that are important in deciding on the order of different types of therapy within one treatment trajectory. The document will guide the therapist in tailoring the treatment trajectory towards the needs of the dyad. The treatment trajectory can consist of EMDR-therapy for the parent, EMDR therapy for the child and NIKA for the parent-child relationship. The guidance document will guide the therapist in deciding on the order of the different therapies.
  Interventions: Behavioral: Guidance document

INTERVENTIONS:
Behavioral: Guidance document — The main intervention of interest is the guidance document, which is explained under 'Arms'. Within the treatment trajectory, that is based on the guidance document, the participants can receive a combination of NIKA, and parent and child can both get EMDR-therapy. The therapies are combined in one treatment trajectory.
  NIKA consists of 5 weekly sessions during which participants are videotaped by a trained therapist. The therapist will provide personalized feedback to the parent, which is focused on reducing disrupted parenting behavior and increasing sensitive parenting behavior. EMDR is a brief trauma therapy (in this trial a maximum of six 90-min sessions for the parent and a maximum of six 60-min sessions for the child) aimed at reducing the negative load of the memories of traumatic events. Both parent and child can receive this therapy. During the weekly sessions, the participant is asked to bring the traumatic event to mind while the therapist provides a distracting task.

SUMMARY:
The goal of this study is to evaluate the effectiveness of an individualized treatment trajectory in which the order of trauma therapy for the parent (Eye movement desensitization and reprocessing (EMDR) therapy), trauma therapy for the child (EMDR therapy) and attachment-based therapy (Dutch short-term intervention for atypical parenting behavior (NIKA)) is tailored towards the complex needs of victimized parents and their young children (4-6 y/o) after domestic violence. The treatment trajectory is based on a guidance document that supports therapists to determine the optimal order of interventions based on a standardized set of factors. The primary goals of this study are:

1. To examine how post-traumatic stress disorder (PTSD)-symptoms of parent and child and parental sensitive and disruptive parenting behavior develop and interact over time, while they follow the individualized treatment trajectory.
2. To test whether the start of the treatment trajectory (e.g. the phase in which parents can receive NIKA and EMDR therapy and their child can receive EMDR therapy) leads to a decrease in disruptive parenting behavior towards the child, an increase in sensitive parenting behavior towards the child, and a decrease in PTSD symptoms of the parent in comparison to the baseline phase.
3. To test whether the start of the treatment trajectory (e.g. the phase in which children can receive EMDR therapy and their parent can receive NIKA and EMDR therapy) leads to a decrease in PTSD symptoms of the child in comparison to the baseline phase.

DETAILED DESCRIPTION:
Rationale:

While the adverse effects of domestic violence on victimized parents and children have been extensively documented, there is still little knowledge on effective intervention approaches for these families. Both parents and children are at risk to develop trauma-related psychopathology after domestic violence. In addition, victimized parents are likely to show disrupted parenting due to their own traumatization (resulting from domestic violence and often also from their own traumatic childhood). This increases the risk for developing a disturbed attachment relationship for the child. Treatment should thus focus at improvement on three levels (parenting behavior and post-traumatic stress (PTSD) symptoms of the parent and the child), and can consist of trauma therapy for parent and child and attachment-based therapy. Since the symptoms in different families may exhibit in different ways, and can interact with each other in a different way, an individualized treatment trajectory that takes these interactions in account may be necessary to allow for maximum symptom reduction.

Study design:

The hypotheses will be tested using a single case experimental design (SCED) study, with a non-concurrent, randomized multiple baseline design. Families who receive treatment after experiencing severe domestic violence will be randomly assigned to a baseline length of 3, 4, 5, 6, 7 or 8 weeks (phase 1), and randomization will occur for two sets of five participants. After the end of the baseline phase, the intervention phase will start, during which dyads will follow an individualized treatment trajectory, consisting of different treatments (phase 2), including EMDR therapy for parent and child to reduce their PTSD symptoms and NIKA to reduce disrupted parenting behavior and increase sensitive parenting behavior. The dyads will participate in weekly appointments throughout the whole duration of the study (both baseline and treatment phase).

Study population:

This study will include 10 parent-child dyads who are residing at a community shelter location in the Netherlands after experiencing domestic violence. Parents with children aged between 4-6 years old will be included if both the parent and the child experience clinically important PTSD-symptoms (based on self-report of the parent). In case that not enough parent-child dyads can be recruited, based on the eligible age range of the child, the age range for the children will be widened, so that children aged between 3-6 years can participate.

ELIGIBILITY:
Inclusion Criteria:

* The non-offending parent and child are residing in a community shelter because of a combination of problems that includes severe domestic violence
* The child is aged between 4-6 years old (if there is more than 1 child in this age range in the family, the parent will be asked to report on the symptoms of both children, and the child with the most severe PTSD symptoms will participate)
* The parent experiences clinically important PTSD-symptoms, as defined by a PCL-score of ≥31
* The child experiences PTSD-symptoms on a clinical level, as defined by a CATS-score of ≥15

Exclusion Criteria:

* Parents with extreme mental health problems (e.g., psychosis) that directly affect their ability to participate in an intervention and require immediate intervention for the parent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in disrupted parenting behavior | Weekly, from the beginning until the end of the research trajectory. The minimum length of the research trajectories (and thus the number of measurements) is 14 weeks, and the maximum duration is 25 weeks.
  Behavioral observations from the dyads are videotaped and coded with the 'Atypical Maternal Behavior Instrument for Assessment and Classification'; AMBIANCE (Bronfman et al., 2009-2014). The AMBIANCE is used to score parental behavior on five dimensions. Based on the scores on these dimensions, an overall score of the level of disruption is determined. The overall score is determined in a range between 1-7, where a higher score indicates more disruptive parenting behavior.
Change in sensitive parenting behavior | Weekly, from the beginning until the end of the research trajectory. The minimum length of the research trajectories (and thus the number of measurements) is 14 weeks, and the maximum duration is 25 weeks.
  Behavioral observations from the dyads are videotaped and coded with the 'Ainsworth Maternal Sensitivity Scale' (Ainsworth et al., 1974). Based on this scale, an overall score is given for the sensitivity of the parent towards the child. The score is given on a range between 1-9, where a higher score indicates a higher level of sensitive behavior of the parent towards the child.
Change in PTSD symptoms of the child | Weekly, from the beginning until the end of the research trajectory. The minimum length of the research trajectories (and thus the number of measurements) is 14 weeks, and the maximum duration is 25 weeks.
  Measured with the 'Child and Adolescent Trauma Screen'; CATS (Sachser et al., 2017). The CATS consists of 16 items, and every item can be scored on a scale of 0-3. Participants can score on a range between 0-48, where a higher score indicates that the child has more PTSD-symptoms.
Change in PTSD symptoms of the parent | Weekly, from the beginning until the end of the research trajectory. The minimum length of the research trajectories (and thus the number of measurements) is 14 weeks, and the maximum duration is 25 weeks.
  Measured with the 'PTSD checklist for DSM-5'; PCL-5 (Boeschoten et al., 2014). The PCL-5 consists of 16 items, and every item can be scored on a scale of 0-4. Participants can score on a range between 0-80, where a higher score indicates that the parent has more PTSD-symptoms.

SECONDARY OUTCOMES:
Quality of life of the child | Weekly, from the beginning until the end of the research trajectory. The minimum length of the research trajectories (and thus the number of measurements) is 14 weeks, and the maximum duration is 25 weeks.
  Measured with 6 questions of the Kiddy-KINDL questionnaire (version for 4-6 year-olds) (Villalonga-Olives et al., 2014). Six positively-formulated items of the Kiddy-KINDL will be used. Every item can be answered on a scale of 1-3. Participants can score on a range between 6-18, where a higher score indicates a better quality of life.
Satisfaction with the treatment trajectory | Only at the end of the research trajectory (post-test). Depending on the total length of the research trajectory, this will be between 14-25 weeks.
  Semi-structured interview with the parent

CONTACTS AND LOCATIONS:
Locations (1):
- HVO Querido, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual participant data and other study materials will be shared upon reasonable request.